CLINICAL TRIAL: NCT05167240
Title: European Society of Hypertension Ambulatory Blood Pressure Monitoring COVID-19 Study
Brief Title: ESH ABPM COVID-19 STUDY
Acronym: ABMP COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Sponsor
Other Study IDs: ESHABPMCOVID-19_01
Record Dates: First submitted 2021-12-21; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Ambulatory Blood Pressure
Keywords: ABPM, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 - will constitute of participants with two repeated ABPM recordings (visits): the second visit performed between 01.04.2020 - 31.03.2021 (i.e., during the COVID-19 pandemic announced by the WHO in 11.03.2020) and the first visit 9-15 months before the second ABPM recording, but not later than 31.12.2019.
- Group 2: Group 2 - will constitute of participants with two repeated ABPM recordings (visits) - both visits performed before the pandemic: the second visit in 01.01.2019 - 31.12.2019 and the first visit 9-15 months before the second.

SUMMARY:
Aim of the study is to determine the impact of the COVID-19 pandemic on blood pressure profiles and variability as assessed by ambulatory blood pressure monitoring (ABPM) through the comparison of ABPM data obtained before and during the COVID-19 lockdown in already treated hypertensive patients

DETAILED DESCRIPTION:
Recruitment for the study will be conducted according to the principles outlined in the Helsinki declaration for investigations in human subjects. The Ethics Committee of each Center must approve the protocol. We will collect clinical data, including office and ambulatory blood pressure of patients with treated arterial hypertension at least 18 years of age.

The study will include two different groups . Group 1 - will constitute of participants with two repeated ABPM recordings (visits): the second visit performed between 01.04.2020 - 31.03.2021 (i.e., during the COVID-19 pandemic announced by the WHO in 11.03.2020) and the first visit 9-15 months before the second ABPM recording, but not later than 31.12.2019.

Group 2 - will constitute of participants with two repeated ABPM recordings (visits) - both visits performed before the pandemic: the second visit in 01.01.2019 - 31.12.2019 and the first visit 9-15 months before the second.

Primary outcome. Difference of changes (deltas) in averaged 24-hour systolic and diastolic BP assessed by ABPM from Visit 1 to Visit 2 between Group 1 and Group 2.

Primary outcome evaluation:

1. Assessment of BP (i.e., average 24hSBP, average 24hDBP) changes (deltas) from values recorded in the year preceding the COVID-19 pandemic to BP (i.e., average 24hSBP, average 24hDBP) values measured during the lockdown (Group 1).
2. Assessment of BP (i.e., average 24hSBP, average 24hDBP) changes (deltas) from values recorded in the pre-pandemic period with 9-15 months' time interval (Group 2).
3. Differences in BP (i.e., average 24hSBP, average 24hDBP) changes (deltas) assessed by ABPM from Visit 1 to Visit 2 between Group 1 and Group 2.

Secondary outcomes:

1. Assessment of BP (i.e., average 24hSBP, average 24hDBP) changes predictors in Group 1 and Group 2.
2. Assessment of differences in averaged Daytime (awake) BP changes assessed by ABPM from Visit 1 to Visit 2 between Group 1 and Group 2.
3. Assessment of differences in averaged Night-time (asleep) BP changes assessed by ABPM from Visit 1 to Visit 2 between Group 1 and Group 2.
4. Assessment of white - coat, masked, and resistant hypertension prevalence in Group 1 and Group 2.
5. Assessment of the extent of asleep BP fall, and dipper/non-dipper phenotypes prevalence in Group 1 and Group 2.
6. Analyses of BP short-term (24hABPM) variability

ELIGIBILITY:
Inclusion Criteria:

1. Pharmacologically treated hypertensive patients.
2. Office systolic, diastolic blood pressure and heart rate available from the day (+/- 1 month) of ABPM recording. If office BP are not available, please provide first BP measurement from ABPM recording.
3. Availability of at least two valid ABPM recordings in 9-15 months interval. a. Group 1 with the second ABPM during the pandemic period: i. First ABPM (visit 1) obtained 9-15 months before the second ABPM recording, but not later than 31.12.2019 ii. Second ABPM (visit 2) obtained during the pandemic period 01.04.2020 - 31.03.2021 b. Group 2 with both ABPM recordings before the pandemic period: i. First ABPM (visit 1) obtained 9-15 months before the Second ABPM ii. Second ABPM (visit 2) obtained between 01.01.2019 - 31.12.2019

Exclusion Criteria:

1. Confirmed secondary hypertension.
2. Hypertension in pregnancy.
3. Device based treatment of hypertension.
4. Development of heart failure, cardiac surgery, myocardial infarction, or cancer between ABPM measurements.
5. Parkinson disease.
6. Alcohol or drug abuse.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will collect clinical data, including office and ambulatory blood pressure of patients with treated arterial hypertension at least 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-06-03 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference of changes in averaged 24-hour systolic and diastolic BP | Visit 2 01.04.2020 - 31.03.2021 and Visit 1 and the first visit 9-15 months before the second ABPM recording, but not later than 31.12.2019
  Difference of changes (deltas) in averaged 24-hour systolic and diastolic BP assessed by ABPM from Visit 1 to Visit 2 between Group 1 and Group 2.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Januszewicz, Prof, Study Chair — National Institute of Cardiology, Warszawa, Poland
Locations (1):
- I Department of Cardiology, Interventional Electrocardiology and Arterial Hypertension, UJ CM, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreutz R, Dobrowolski P, Prejbisz A, Algharably EAE, Bilo G, Creutzig F, Grassi G, Kotsis V, Lovic D, Lurbe E, Modesti PA, Pappaccogli M, Parati G, Persu A, Polonia J, Rajzer M, de Timary P, Weber T, Weisser B, Tsioufis K, Mancia G, Januszewicz A; European Society of Hypertension COVID-19 Task Force Review. Lifestyle, psychological, socioeconomic and environmental factors and their impact on hypertension during the coronavirus disease 2019 pandemic. J Hypertens. 2021 Jun 1;39(6):1077-1089. doi: 10.1097/HJH.0000000000002770. PMID 33395152
- [Background] Pecanha T, Goessler KF, Roschel H, Gualano B. Social isolation during the COVID-19 pandemic can increase physical inactivity and the global burden of cardiovascular disease. Am J Physiol Heart Circ Physiol. 2020 Jun 1;318(6):H1441-H1446. doi: 10.1152/ajpheart.00268.2020. Epub 2020 May 15. PMID 32412779
- [Background] The corona-virus disease 2019 pandemic compromised routine care for hypertension: a survey conducted among excellence centers of the European Society of Hypertension. J Hypertens. 2021 Jan;39(1):190-195. doi: 10.1097/HJH.0000000000002703. PMID 33273364
- [Background] Kreutz R, Algharably EAE, Azizi M, Dobrowolski P, Guzik T, Januszewicz A, Persu A, Prejbisz A, Riemer TG, Wang JG, Burnier M. Hypertension, the renin-angiotensin system, and the risk of lower respiratory tract infections and lung injury: implications for COVID-19. Cardiovasc Res. 2020 Aug 1;116(10):1688-1699. doi: 10.1093/cvr/cvaa097. PMID 32293003
- [Background] Pengo MF, Albini F, Guglielmi G, Mollica C, Soranna D, Zambra G, Zambon A, Bilo G, Parati G. Home blood pressure during COVID-19-related lockdown in patients with hypertension. Eur J Prev Cardiol. 2022 Mar 25;29(3):e94-e96. doi: 10.1093/eurjpc/zwab010. No abstract available. PMID 33899916
- [Background] Stergiou GS, Palatini P, Parati G, O'Brien E, Januszewicz A, Lurbe E, Persu A, Mancia G, Kreutz R; European Society of Hypertension Council and the European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. 2021 European Society of Hypertension practice guidelines for office and out-of-office blood pressure measurement. J Hypertens. 2021 Jul 1;39(7):1293-1302. doi: 10.1097/HJH.0000000000002843. No abstract available. PMID 33710173
- [Background] Hoshide S, Kario K. Morning Surge in Blood Pressure and Stroke Events in a Large Modern Ambulatory Blood Pressure Monitoring Cohort: Results of the JAMP Study. Hypertension. 2021 Sep;78(3):894-896. doi: 10.1161/HYPERTENSIONAHA.121.17547. Epub 2021 Jul 26. No abstract available. PMID 34304583
- [Background] Mena L, Pintos S, Queipo NV, Aizpurua JA, Maestre G, Sulbaran T. A reliable index for the prognostic significance of blood pressure variability. J Hypertens. 2005 Mar;23(3):505-11. doi: 10.1097/01.hjh.0000160205.81652.5a. PMID 15716690
- [Background] Bilo G, Giglio A, Styczkiewicz K, Caldara G, Maronati A, Kawecka-Jaszcz K, Mancia G, Parati G. A new method for assessing 24-h blood pressure variability after excluding the contribution of nocturnal blood pressure fall. J Hypertens. 2007 Oct;25(10):2058-66. doi: 10.1097/HJH.0b013e32829c6a60. PMID 17885548